CLINICAL TRIAL: NCT02491294
Title: Cooking With Kids 2.0: Plus Parents and Play
Brief Title: Fuel for Fun: Cooking With Kids Plus Parents and Play
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Penn State University (Other); Poudre School District (Unknown); Thompson School District (Unknown); Rochester Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 12-3278H
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Obesity
Keywords: School; Family; Fruit and Vegetables; Cooking; Physical Activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- School Only (Experimental): Students whose schools are randomized to this condition only receive the classroom, cafeteria and SPARK active recess components
  Interventions: Behavioral: School
- School + Family (Experimental): Students whose schools are randomized to this condition receive the classroom, cafeteria and SPARK active recess components and the family component (family nights, parent blog and action packs)
  Interventions: Behavioral: School; Behavioral: Family
- School + About Eating (Experimental): Students whose schools are randomized to this condition only receive the classroom, cafeteria and SPARK active recess components and their parents are invited to participate in the online 6 lesson About Eating program.
  Interventions: Behavioral: School; Behavioral: About Eating
- School + Family + About Eating (Experimental): students whose schools are randomized to this condition receive the classroom, cafeteria and SPARK active recess components and the family component (family nights, parent blog and action packs) and their parents are invited to participate in the online 6 lesson About Eating program.
  Interventions: Behavioral: School; Behavioral: Family; Behavioral: About Eating
- Control (No Intervention): students and their parents in all schools during cohort 1 and 4 (and Ponderosa students in cohort 3) are tested but provided no intervention

INTERVENTIONS:
Behavioral: School — students receive Cooking With Kids (CWK) - Colorado cooking & tasting lessons, SPARK active recess, and Cafeteria Connections
  Arms: School + About Eating; School + Family; School + Family + About Eating; School Only
Behavioral: Family — students receive the FFF family component - family nights, parent blog, and action packs that go home after each CWK-Colorado lesson
  Arms: School + Family; School + Family + About Eating
Behavioral: About Eating — parents who completed the parent survey are invited to access the 6 lesson online About Eating program
  Arms: School + About Eating; School + Family + About Eating

SUMMARY:
Fuel for Fun: Cooking with Kids Plus Parents and Play (FFF), is an integrated research, extension, and education project targeting 4th grade students. Its long-term goal of reducing the risk of childhood obesity will be addressed by promoting healthful food and activity environments, policies and behaviors through: 1) building and testing the efficacy of a 4th grade comprehensive school- and family-based intervention, 2) applying it to an after-school setting to broaden its reach, and, 3) disseminating both versions through outreach.

DETAILED DESCRIPTION:
Fuel for Fun: Cooking with Kids Plus Parents and Play (FFF) is based on existing, evidence-based components: the experiential Cooking with Kids curriculum, the SPARK Active Recreation program; principles of behavioral economics in school cafeterias and homes; the online About Eating 5-lesson module based on eating competence concepts, and a family-based FFF component specifically designed for this intervention.

Each component addresses policy and environment in addition to behavior change at school and home. The main research project - school-based FFF - will be implemented in 8 low-to-moderate income schools for two years using an asynchronous design that allows for assessment of the school-based program alone and in combination with both parent programs. Changes in fruit and vegetable intake (measured by self-report, cafeteria plate waste) and activity levels (measured by self-report and accelerometry) are primary outcomes, with measured BMI as a secondary outcome. Subsequent studies will involve the development of an after-school version and adoption of FFF by other districts.

University students will gain valuable research experience and school and Extension educators will receive important childhood obesity prevention training. The project's long term goal is consistent with the United States Department of Agriculture (USDA) goal of improving the nation's nutrition and health by promoting the development of healthy eating and activity habits in children.

ELIGIBILITY:
Inclusion Criteria:

* all students enrolled in participating classrooms are invited to participate

Exclusion Criteria:

* none

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2640 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Consumption at School Lunch | assessed 4 times each 9-month school year; once prior to intervention beginning (i.e., September), approximately 10 weeks and then 20 weeks later, and finally once after the intervention ends (i.e., May).
  using observation and digital photography we will assess student selection and consumption of fruits and vegetables during school lunch; measured at the grade level
Change in Student Activity Level | assessed 3 times over 1 year; initially prior to the intervention beginning (i.e., September), a 2nd time once the intervention ends (i.e., May), and then again at the beginning of the following school year (i.e., September)
  Using accelerometers, we will assess a week of activity; 3 of 8 participating schools have been randomized to participate in this data collection

SECONDARY OUTCOMES:
Body Mass Index | assessed 3 times over 1 year; initially prior to the intervention beginning (i.e., September), a 2nd time once the intervention ends (i.e., May), and then again at the beginning of the following school year (i.e., September)
  using a standard protocol, we will measure height and weight of all participating students and then calculate BMI z-scores

CONTACTS AND LOCATIONS:
Locations (1):
- Leslie Cunningham-Sabo, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Once all data has been collected, analyzed and published we plan to explore how to share de-identified accelerometry data for children and adults.

REFERENCES:
- [Derived] Cunningham-Sabo L, Lohse B, Clifford J, Burg A, Nigg C. Fuel for Fun Process Evaluation Reveals Strong Implementation and Approval with Varied Parent Engagement. J Nutr Educ Behav. 2023 Jan;55(1):16-29. doi: 10.1016/j.jneb.2022.08.001. PMID 36621265
- [Derived] Lohse B, Faulring K, Mitchell DC, Cunningham-Sabo L. A Definition of "Regular Meals" Driven by Dietary Quality Supports a Pragmatic Schedule. Nutrients. 2020 Sep 1;12(9):2667. doi: 10.3390/nu12092667. PMID 32882978
- [Derived] Cunningham-Sabo L, Lohse B, Smith S, Browning R, Strutz E, Nigg C, Balgopal M, Kelly K, Ruder E. Fuel for Fun: a cluster-randomized controlled study of cooking skills, eating behaviors, and physical activity of 4th graders and their families. BMC Public Health. 2016 May 26;16:444. doi: 10.1186/s12889-016-3118-6. PMID 27230565